CLINICAL TRIAL: NCT06600490
Title: Nationwide Utilization of Danish Government Electronic Letter System for Confirming the Effectiveness of Behavioral Nudges in Increasing InFLUenza Vaccine Uptake Among Adults With Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUDGE-FLU-CHRONIC-2
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza; Behavior and Behavior Mechanisms
Keywords: Influenza; Vaccination; Nudging; Behavioral Science; Randomized Trial; Registry
MeSH Terms: conditions — Influenza, Human; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Usual Care (No Intervention): No letter
- Standard Letter (Experimental): This group will receive a standard letter on the benefits of influenza vaccination without behavioral economic enhancement
  Interventions: Behavioral: Behavioral Economic Principles
- Repeated Letter (Experimental): The standard letter sent out two times instead of once
  Interventions: Behavioral: Behavioral Economic Principles
- Cardiovascular Gain-Framing Letter (Experimental): Text added to the standard letter highlighting potential cardiovascular benefits of influenza vaccination
  Interventions: Behavioral: Behavioral Economic Principles
- Repeated Cardiovascular Gain-Framing Letter (Experimental): The cardiovascular gain-framing letter sent out two times instead of once
  Interventions: Behavioral: Behavioral Economic Principles
- Respiratory Gain-Framing Letter (Experimental): Text added to the standard letter highlighting potential respiratory disease-related benefits of influenza vaccination
  Interventions: Behavioral: Behavioral Economic Principles
- Implementation Intention Prompt Letter (Experimental): Implementation intention prompt added to the standard letter
  Interventions: Behavioral: Behavioral Economic Principles

INTERVENTIONS:
Behavioral: Behavioral Economic Principles — The control arm will receive no letter to reflect the background vaccination uptake. Intervention arms will test the effects of different letters developed using behavioral economic principles.
  Arms: Cardiovascular Gain-Framing Letter; Implementation Intention Prompt Letter; Repeated Cardiovascular Gain-Framing Letter; Repeated Letter; Respiratory Gain-Framing Letter; Standard Letter

SUMMARY:
In randomized clinical trials and observational studies, influenza vaccination has been shown to be effective in reducing influenza-related illness, hospitalizations, cardiovascular events, and mortality in select populations. However, the real-world effectiveness of influenza vaccination is limited by its uptake. Conducted during the 2023/2024 influenza season, the first NUDGE-FLU-CHRONIC trial demonstrated the effectiveness of behavioral nudging letters in increasing influenza vaccination rates among adults aged 18-64 years with chronic diseases in Denmark. This present study will once again investigate whether digital behavioral nudges delivered via the official, mandatory Danish electronic letter system can increase influenza vaccine uptake among adults aged 18-64 years with chronic diseases including whether the effectiveness of the previously successful strategies can be confirmed during a subsequent influenza season.

DETAILED DESCRIPTION:
The study is a prospective, randomized, open-label implementation trial. The study population will consist of persons aged 18-64 years identified as eligible for free-of-charge influenza vaccination due to a chronic condition. Subjects will be identified through Danish nationwide health registries using codes from the International Classification of Diseases, 10th revision (ICD-10). Individuals will be randomized to 1 of 7 arms (1 usual care arm and 6 intervention arms) with each testing different nudging strategies employing various behavioural economic principles. The interventions will be delivered through the official, mandatory Danish electronic letter system. All subject data will be retrieved from the Danish nationwide registries with the exception of information on intervention allocation. Endpoints will be retrieved at prespecified dates using prespecified search algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64 years
2. Must be registered in the Danish nationwide registries as meeting at least one of the following eligibility criteria for free-of-charge influenza vaccination in the Danish public health system:

   1. Chronic lung disease
   2. Chronic cardiovascular disease other than hypertension
   3. Type 1 or type 2 diabetes mellitus
   4. Congenital or acquired immunodeficiency
   5. Impaired breathing due to muscular weakness
   6. Chronic renal or hepatic insufficiency
   7. Other chronic conditions with an increased risk of severe influenza as determined by the treating physician
3. Access to the official, mandatory Danish electronic mailbox system

Exclusion Criteria:

None

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308978 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received an influenza vaccine | Up to 3 months

SECONDARY OUTCOMES:
Time from intervention delivery to influenza vaccination | Up to 3 months

OTHER OUTCOMES:
Number of participants with laboratory-confirmed influenza | Up to 8 months
Number of participants with a hospitalization for influenza or pneumonia | Up to 8 months
Number of participants with a hospitalization for any respiratory disease | Up to 8 months
Number of participants with a hospitalization for any cardio-respiratory disease | Up to 8 months
Number of participants with a hospitalization for any cardiovascular disease | Up to 8 months
Number of participants with any hospitalization | Up to 8 months
Total number of hospitalizations (first and recurrent) | Up to 8 months
All-cause mortality | Up to 8 months
Composite of incident heart failure, heart failure hospitalization, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, stroke, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, coronary revascularization, stroke, or cardiovascular death | Up to 8 months
Number of participants with incident heart failure or heart failure hospitalization | Up to 8 months
Total number of heart failure events (incident heart failure and first and recurrent heart failure hospitalizations) | Up to 8 months
Cardiovascular death | Up to 8 months
Number of participants with myocardial infarction | Up to 8 months
Number of participants with coronary revascularization | Up to 3 months
Number of participants with stroke | Up to 8 months
Number of participants with incident atrial fibrillation or atrial fibrillation hospitalization | Up to 8 months
Number of contacts to general practitioner (excluding vaccination visit) | Up to 8 months
Number of participants with laboratory-confirmed COVID-19 | Up to 8 months
Number of participants with a hospitalization for COVID-19 | Up to 8 months
Number of participants who received a COVID-19 vaccine | Up to 3 months
Number of participants who filled a prescription for any guideline-directed medical therapy for heart failure | Up to 8 months
Total number of filled prescriptions for guideline-directed medical therapy for heart failure | Up to 8 months
Number of participants who filled a prescription for a sodium-glucose cotransporter 2 inhibitor or glucagon-like peptide 1 receptor agonist | Up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Principal Investigator — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.

REFERENCES:
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Modin D, Claggett BL, Janstrup KH, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Krause TG, Biering-Sorensen T. Digital Nudges to Increase Influenza Vaccination in Patients with Chronic Diseases. NEJM Evid. 2026 Jan;5(1):EVIDoa2500265. doi: 10.1056/EVIDoa2500265. Epub 2025 Nov 10. PMID 41213006